CLINICAL TRIAL: NCT03156049
Title: Sphenopalatine Ganglion Block Versus Occiptal Nerve Block in Treatment of Postduarl Puncture Headache
Brief Title: Sphenopalatine Ganglion Block Versus Occiptal Nerve Block in Treatment of Post Dural Puncture Headache
Acronym: PDPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, Assisstant professor in anesthesia and intensive care, Faculty of medicine, Assiut university, Egypt., Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17200061
Record Dates: First submitted 2017-05-14; First posted 2017-05-17 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Headache
MeSH Terms: conditions — Headache | interventions — Sphenopalatine Ganglion Block

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sphenopalatine block (Active Comparator): patients will receive bilateral sphenopalatine ganglion block using 3ml mixture of 2ml 2% lidocaine plus 1ml dexamethasone 4mg (on each nostril).
  Interventions: Procedure: Sphenopalatine block
- Greater occipital nerve block (Active Comparator): patients will receive bilateral greater occipital nerve block using a mixture of 3ml of 2ml 2% lidocaine plus 1ml dexamethasone 4mg (on each side of the occipital region).
  Interventions: Procedure: Greater occipital nerve block

INTERVENTIONS:
Procedure: Sphenopalatine block — patients will receive bilateral sphenopalatine ganglion block using 3ml mixture of 2ml 2% lidocaine plus 1ml dexamethasone 4mg (on each nostril).
  Other Names: SPGB
  Arms: Sphenopalatine block
Procedure: Greater occipital nerve block — patients will receive bilateral greater occipital nerve block using a mixture of 3ml of 2ml 2% lidocaine plus 1ml dexamethasone 4mg (on each side of the occipital region).
  Other Names: GONB
  Arms: Greater occipital nerve block

SUMMARY:
Postdural puncture headache (PDPH) is a common complication associated with neuraxial anesthesia and diagnostic lumbar puncture (LP). PDPH is defined as a bilateral headache that develops within 7 days and disappears within 14 days after the dural puncture with a distinct postural quality. PDPH causes significant short-term disability, prevents ambulation and care of the newborn (in obstetrics), and results in a prolonged hospital stay.

DETAILED DESCRIPTION:
The sphenopalatine ganglion (SPG) is an extra-cranial neural structure located in the pterygopalatine fossa that has both sympathetic and parasympathetic components as well as somatic sensory roots. The trans-nasal approach is a low risk, noninvasive technique that is easily performed and could potentially be beneficial in the treatment of PDPH through blocking the parasympathetic ﬂow to the cerebral vasculature through the sphenopalatine ganglion which will allow the cerebral vessels to return to normal diameter and thus relieve the headache.

The greater occipital nerve contains sensory fibers from C2 and C3 segments of medulla spinals. It arises from the dorsal ramus of C2 segment, contains a thin branch from C3 segment, and innerves the medial aspect of posterior scalp up to the anterior aspect of vertex. Greater occipital nerve block (GONB) inhibits the pain sensation of this region.

There is some evidence to suggest the effectiveness of GONB in the management of PDPH. Nowadays, guidelines for the management of PDPH were modified and included GONB as a part of standard management of PDPH.

* Dexamethasone possess potent antiinflammatory and immunosuppressive actions by inhibiting cytokine-mediated pathways.
* Many providers believe that the local anesthetic produces the rapid onset of headache relief, like an abortive agent, and that the locally acting steroid produces the preventive like action of up to 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

ASA I-II Patients undergoing elective cesarean section requiring spinal anesthesia, who developed PDPH during hospitalization or within days of the intrathecal block.

Exclusion Criteria:

* Patient refusal.
* Any contraindication to regional block (coagulopathy or anticoagulant therapy).
* Local scalp infection.
* Nasal polyp, trauma, septal deviation or any nasal pathology.
* Allergy to local anesthetics.
* Pregnancy induced hypertension.
* History of major psychiatric disorders.
* Chronic headache.
* Substance abuse.
* Current opioid use.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Numeric rating pain score | from intervention up to 24 hours
  pain score

SECONDARY OUTCOMES:
Numeric rating pain score for headache. | from intervention up to 24 hours
  pain score
Analgesic consumption | from intervention up to 24 hours
  The total dose of analgesics.

CONTACTS AND LOCATIONS:
Overall Officials: Hala Abdel-Ghaffar, MD, Principal Investigator — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Assiut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No